CLINICAL TRIAL: NCT01189513
Title: A Phase I Evaluation of SCH 900105 With Correlative Tissue Studies in the Treatment of Adult Patients With Recurrent Glioblastoma
Brief Title: SCH-900105 in Recurrent Glioblastoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0576
Record Dates: First submitted 2010-08-25; First posted 2010-08-26 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Glioblastoma
Keywords: Recurrent Glioblastoma; Gliosarcoma; SCH 900105
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — ficlatuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SCH 900105 (Experimental): 10 mg/kg intravenous Days 1, 8 and 15 of 30 day cycle.
  Interventions: Drug: SCH 900105

INTERVENTIONS:
Drug: SCH 900105 — 10 mg/kg by vein every week on days 1, 8 and 15 of a 30 day cycle.

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of SCH 900105 that can be given to patients with glioblastoma before surgery. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
The Study Drug:

SCH 900105 is designed to block the activity of one of the tumor-causing proteins responsible for the development and uncontrolled growth of tumor cells and the formation of new blood vessels. This may result in shrinking or stopping tumor growth.

You will need to take SCH 900105 for 14 days before surgery. If the doctor decides there is a risk from the delay of surgery, you will not be able to take part in this study.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a dose level of SCH 900105 based on when you joined this study. Up to 3 dose levels (Dose Levels 0, 1, and 2) of SCH 900105 will be tested before surgery. Three (3) participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level (Dose Level 0). Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of SCH 900105 is found.

No matter what dose level you are assigned before surgery, all participants will receive Dose Level 1 of SCH 900105 after surgery.

The amount of study drug you receive may change if you experience side effects. If at any time you experience any intolerable side effects, tell the study doctor right away.

Study Drug Administration:

Cycle 1 will be 30 days and each following cycle will be 28 days.

If you are assigned to Dose Levels 0 or 2, you will receive SCH 900105 by vein over about 1 hour on Days 1, 8, and 15 of Cycle 1.

If you are assigned to Dose Level 1, you will receive SCH 900105 by vein over about 1 hour on Days 1 and 15 of Cycle 1.

As a part of standard of care, you will have a surgery to remove the regrown tumor on Day 16 of Cycle 1. You will sign a separate consent for this surgery, which will describe the procedure and its risks in detail.

You will not receive SCH 900105 for about 2 weeks after surgery. After 2 weeks, you will receive SCH 900105 by vein on Days 1 and 15 of each cycle (Cycles 2 and beyond).

Study Visits:

At every visit, you will be asked about any drugs you may be taking and if you have experienced any side effects.

On Days 1, 8, 15, and 22 of Cycle 1, blood (about 2 teaspoons) will be drawn for routine tests.

On Day 17 of Cycle 1, you will have an MRI scan to check the status of the disease.

On Day 1 of Cycles 2 and beyond:

* Your complete medical history will be recorded. You will have a physical exam, including measurement of your weight and vital signs.
* You will have a neurological exam.
* Your performance status will be recorded.
* Blood (about 2 teaspoons) will be drawn for routine tests.

On Day 15 of Cycles 2 and beyond, blood (about 2 teaspoons) will be drawn for routine tests.

On Day 1 of every other cycle starting Cycle 3 (Cycles 3, 5, 7, and so on), you will have an MRI scan to check the status of the disease.

Pharmacokinetic (PK) and Biomarker Tests:

Extra blood will be drawn for PK testing and biomarker testing. PK testing measures the amount of study drug in the body at different time points. These tests are for research only.

Blood (about 1 teaspoon each time) will be drawn during the following times for PK testing:

* On Day 1 of Cycle 1, blood will be drawn 4 times.
* On Day 15 of Cycle 1, blood will be drawn 3 times.
* On Days 16, 17, and 19 of Cycle 1, blood will be drawn 1 time.
* On Day 1 of Cycles 2 and beyond, blood will be drawn 1 time.
* At 45 and 60 days after the last dose of SCH 900105, blood will be drawn 1 time.
* If you are assigned to Dose Levels 0 or 2, blood will also be drawn 2 times on Day 8 of Cycle 1.

Blood (about 2 teaspoons each time) will be drawn during the following times for biomarker testing:

* On Days 1 and 15 of Cycle 1, blood will be drawn 1 time.
* On Day 1 of Cycles 2 and beyond, blood will be drawn 1 time.
* If you are assigned to Dose Levels 0 or 2, blood will also be drawn 1 time on Day 8 of Cycle 1.

Leftover tumor tissue (removed during your surgery on Day 16 of Cycle 1) will be collected and used for PK tests and biomarker tests.

Length of Study:

You may continue receiving SCH 900105 for as long as you are benefitting. You will be taken off study if the disease gets worse or you experience intolerable side effects.

This is an investigational study. SCH 900105 is not FDA approved or commercially available. At this time, SCH 900105 is only being used in research.

Up to 21 patients will be enrolled in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have a diagnosis of supratentorial glioblastoma or gliosarcoma by pathology review after initial tumor resection and who have radiographic evidence of recurrent tumor.
2. Eligibility will be restricted to patients in whom the clinical decision has been made to perform surgery at recurrence for symptom relief or for cytoreduction. Due to the requirement that SCH 900105 treatment will be given for 15 days prior to surgery, only patients who are determined to be not at risk from this delay in the best clinical judgment of the neurosurgeon, the treating neuro-oncologist and the study chair will be eligible for entry into the study.
3. (2. continued) Patients who are in poor clinical condition as defined by Karnofsky performance status (KPS) or have progressive symptoms necessitating urgent surgery will be excluded from this study.
4. Patients must have enhancing disease on the MRI scan sufficient to provide tissue samples for pathological diagnosis & correlative studies AND if the surgical plan includes resection of this part of the tumor. Patients with radiologically evident areas of tumor necrosis will be eligible for entry into this study if there is sufficient non-necrotic tumor to permit tissue correlative studies. The study chair will make a determination with the help of the treating physician, neuro-radiologist and neurosurgeon whether a particular patient fulfils the radiological requirements for study entry.
5. Patients must have failed prior radiation therapy and must have an interval of greater than or equal to 12 weeks (84 Days) from the completion of radiation therapy to study entry.
6. Patients may have had treatment for no more than 3 prior relapses. Relapse is defined as progression following initial therapy (i.e. radiation +/- chemo if that was used as initial therapy). The intent therefore is that patients had no more than 4 prior therapies (initial and treatment for 3 relapses). For patients who had prior therapy for a low-grade glioma, a prior surgical diagnosis of a high-grade glioma will be considered the first relapse.
7. Patients must have recovered from the toxic effects of prior therapy at the time of initiation of the study drug: 4 weeks from any investigational agents, two weeks from vincristine, 6 weeks from nitrosoureas, 3 weeks from procarbazine administration, 3 weeks for temozolomide, 4 weeks for carboplatin, and 1 week for non-cytotoxic agents, e.g., interferon, tamoxifen, cis-retinoic acid, etc. (radiosensitizer does not count). Prior anti-angiogenic therapy is not allowed. For patients who have undergone radiation therapy (XRT), at least 12 weeks should have elapsed since completion of XRT.
8. Patients must be equal to or greater than 18 years of age.
9. All patients must sign an informed consent indicating that they are aware of the investigational nature of this study. Patients must have signed an authorization for the release of their protected health information.
10. Patients must have adequate bone marrow function (absolute granulocyte count >/= 1,500 and platelet count >/= 100,000), normal coagulation profile (PT/PTT), adequate liver function (SGPT, SGOT, and alkaline phosphatase </= 2.5 times normal and bilirubin < 1.5 mg/dL), adequate renal function (BUN or creatinine </= 1.5 times institutional normal) and institutional normal serum amylase within 14 days prior to starting therapy.
11. Patients must have a Karnofsky performance status (KPS) of >/= 60.
12. All patients (men and women) of childbearing potential must agree to use adequate birth control (barrier methods) during and for 1 month after participation in this study.
13. Women of childbearing potential must have a negative Beta Human Chorionic Gonadotropin(B-HCG) pregnancy test documented within 14 days prior to registration.
14. This study was designed to include women and minorities, but was not designed to measure differences of intervention effects. Males and females will be recruited with no preference to gender.
15. Archived paraffin embedded tissue (15 unstained slides) must be available for confirmation of tumor diagnosis and correlative studies prior to receiving the first dose of SCH 900105.

Exclusion Criteria:

1. Patients who have been previously treated with c-Met inhibitors are ineligible for this study.
2. Patients must not have any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy.
3. Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years are ineligible.
4. Patients must not have active infection or with a fever >/= 38.5°C within 3 days prior to the first dose of SCH 900105.
5. Patients must not be pregnant/breast feeding during and for 1 month after participation in this study.
6. Patients must not have any disease that will obscure toxicity or dangerously alter drug metabolism.
7. Patients on full-dose anticoagulants (e.g., warfarin, low molecular weight heparin) for the treatment of deep vein thrombosis(DVT), pulmonary emboli (PE), atrial fibrillation, myocardial infarction, or any other thromboembolic event are not eligible.
8. No exclusion to this study will be based on race. Minorities will actively be recruited to participate. The malignant glioma patient population treated at MDACC over the past year is as follows: American Indian or Alaskan Native - 0; Asian or Pacific Islander - <2%; Black, not of Hispanic Origin - 3%; Hispanic - 6%; White, not of Hispanic Origin - 88%; Other or Unknown - 2%; Total - 100%
9. The safety profile of SCH 900105 was not established in the pediatric population, Patients under age 18 will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 30 days for Cycle 1, and every 28 days for following cycles
  MTD of SCH 900105 defined as the dose level prior to that resulting in dose limiting toxicity (DLT i.e., the dose level at which no more than 1 out of 6 subjects experiences). DLT).

CONTACTS AND LOCATIONS:
Overall Officials: John DeGroot, MD, Principal Investigator — UT MD Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org